CLINICAL TRIAL: NCT03983122
Title: Long Term Outcomes of Laparoscopic Sleeve Gastrectomy: First Five Years' Results of a Single Center From a Developing Country
Brief Title: Outcomes of Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Hakan Seyit, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BakirkoySKGeneralSurgery
Record Dates: First submitted 2019-05-25; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Bariatric Surgery Candidate; Laparoscopic Sleeve Gastrectomy; Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients who undergo laparoscopic sleeve gastrectomy
  Interventions: Procedure: Laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Each procedure will be completed with laparoscopy with five trocars. A 36F bougie will used to calibrate the volume of the remnant stomach. Linear gastrectomy will begin 2 cm proximal of the pylor and will continue until the gastroesophageal junction. According to the intraoperative decision and experience of the surgeon, endoscopic clips would be used to ensure hemostasis of the stapler line.

SUMMARY:
The aim of this study is to assess 5 year long-term outcomes of laparoscopic sleeve gastrectomy emphasizing weight loss and modification of comorbidities such as type 2 diabetes mellitus, hypertension and gastroesophageal reflux disease from a developing country, Turkey. Prospectively-collected patient data will retrospectively reviewed. To measure the efficacy of the procedure, we will calculate the excess weight loss percentage (EWL %). Effective weight loss after LSG will accepted as more than 50%. The changes in the status of the type 2 diabetes mellitus, hypertension, gastroesophageal reflux disease will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were, patients between 18 to 65 years old, initial body mass index (BMI) 40 kg/m2 or BMI of 35 kg/m2 in the presence of additional comorbidity and failure of conservative treatment for 2 years.

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Weight loss | 5 years
  Weight loss after surgery

SECONDARY OUTCOMES:
Remision of comorbid diseases | 5 years
  The pharmacological treatment status of comorbidities related to obesity of type 2 diabetes (T2DM) and hypertension and gastroesophageal reflux will be observed with questions about "did it stop after surgery (improvement), did the dose or number of medications used reduce (resolution), or were there no changes?"